CLINICAL TRIAL: NCT05966701
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Dose Escalation Phase I Clinical Study of Humanized Monoclonal Antibody Injection (SSGJ-613) in Healthy Adult Chinese Subjects
Brief Title: The MAD Study of SSGJ-613 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-613-HH-I-02
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Arthritis, Gouty
MeSH Terms: conditions — Arthritis, Gouty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSGJ-613 (Experimental): SSGJ-613，SC
  Interventions: Drug: SSGJ-613
- Placebo (Placebo Comparator): Placebo, SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SSGJ-613 — SSGJ-613 subcutaneous injection.
  Arms: SSGJ-613
Drug: Placebo — Placebo subcutaneous injection.
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of SSGJ-613 after multiple subcutaneous injections in healthy subjects.

DETAILED DESCRIPTION:
The purposes of this study are to evaluate the safety and tolerability, PK characteristics and immunogenicity of SSGJ-613 after multiple subcutaneous injections in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese healthy participants, male or female, aged 18 to 45 (including both ends)
2. The body mass index (BMI) is in the range of 19.0~28.0 kg•m-2 (including both ends), and the weight of men is generally not less than 50kg, while the women is generally not less than 45kg
3. Participants should fully understand the purpose, nature, methods and possible adverse reactions of the trial, volunteer to participate in the trial and sign the informed consent

Exclusion Criteria:

1. Those who are allergic to the study drug and any of its excipients. Subjects who have a history of allergy to monoclonal antibodies
2. Subjects who have or are currently suffering from any serious clinical diseases before screening,
3. Abnormal vital signs or abnormal ECGor physical examination are clinically significant
4. Clinical laboratory examinations found to be abnormal and have clinical significance
5. Positive for Hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HbcAb), anti- Hepatitis C virus antibodies (HCV), or anti-human immunodeficiency virus (HIV)
6. Alcoholics or frequent drinkers within 3 months before the trial, drinking more than 14 units per week (1 unit alcohol ≈360 mL beer or 45 mL spirits or 150 mL wine), or those who have a positive alcohol breath test (screening period or baseline period) or couldn't prohibit alcohol during the trial
7. Drug abusers or those who have used soft drugs (such as marijuana) within 3 months or took hard drugs (such as cocaine, phencyclidine, etc.) within 1 year before the trial, or have positive drug abuse screening
8. Has taken any prescription medicine, non-prescription medicine, Chinese patent medicine within 2 weeks before administration
9. Has known or suspected pregnancy or lactation
10. Subjects who are unsuited to the study for any reason, judged by the investigators

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs), measurement of vital signs，physical examination，electrocardiogram and laboratory tests at each visit. | Up to Day 174
  The incidence and severity of treatment emergent adverse event (TEAE), including Serious Adverse Event (SAE), as well as clinical symptoms, and any abnormalities of vital signs, physical examinations，electrocardiogram，laboratory tests and, etc..

SECONDARY OUTCOMES:
SSGJ-613 Concentration in Serum | Up to Day 174
  The concentration of SSGJ-613 in Serum.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghong Zhou, BS, Study Director — Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd.; Qian Chen, PhD, Principal Investigator — Shanghai Xuhui District Central Hospital
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No